CLINICAL TRIAL: NCT07097649
Title: Investigation of the Effects of Lateral Wedge Textured Insoles on Balance, Physical Performance, and Plantar Pressure Distribution in Older Adults With Medial Knee Osteoarthritis
Brief Title: Effects of Textured Insoles on Balance, Physical Performance, and Plantar Pressure in Older Adults With Knee Osteoarthritis
Acronym: TIKOA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Nur Turkmen (Other)
Responsible Party: Sponsor-Investigator, Esra Nur Turkmen, PhD Lecturer, Principal Investigator - Department of Physiotherapy and Rehabilitation, KSÜ, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHU-TEXTINSOLE-2025-01
Record Dates: First submitted 2025-07-18; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: Medial Compartment Knee Osteoarthritis; Textured Insoles; Balance; Plantar Pressure; Physical Performance
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel arms: the intervention group will receive textured lateral wedge insoles, and the control group will receive flat lateral wedge insoles without texture.
  Both groups will wear the insoles in their daily footwear for 4 weeks. All participants will be assessed using standardized protocols covering balance, plantar pressure distribution, physical performance, and biomechanical parameters, through objective measurement systems.
Masking Description: No parties were masked due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Textured insoles group (Experimental): Participants will use textured insoles for 8 weeks.
  Interventions: Device: Textured lateral wedge insole
- Lateral wedge flat insoles group (Active Comparator): The researchers will use flat insoles with lateral wedges for 8 weeks.
  Interventions: Device: Use of lateral wedge flat insole

INTERVENTIONS:
Device: Textured lateral wedge insole — Participants in the experimental group will wear custom-designed textured lateral wedge insoles made from EVA material. These insoles incorporate lateral wedging to offload the medial knee compartment and a textured surface to enhance plantar sensory input. Participants will use the insoles during daily activities for a period of 8 weeks, with no additional intervention or exercise protocol.
  Other Names: Lateral wedge textured insole
  Arms: Textured insoles group
Device: Use of lateral wedge flat insole — Participants in this arm will use a customized lateral wedge flat insole with the same lateral inclination as the experimental insole but without any textured surface. This design allows for controlling the mechanical effect of the wedge while eliminating additional sensory stimulation.
  Arms: Lateral wedge flat insoles group

SUMMARY:
This study aims to investigate the effects of textured insoles on balance, physical performance, and plantar pressure distribution in older adults with medial compartment knee osteoarthritis. Participants will be randomly assigned to two groups: the intervention group will receive textured insoles, while the control group will receive flat insoles without texture. Both groups will use their respective insoles for 4 weeks in their daily life. The study includes pre- and post-intervention assessments using balance platforms, functional performance tests (such as the Timed Up and Go, 30-second Chair Stand Test, and Step Test), and plantar pressure analysis. This randomized controlled study is designed to evaluate the effectiveness of textured insoles as a non-invasive and easily applicable rehabilitation method in improving balance and pressure distribution in elderly individuals with knee osteoarthritis.

DETAILED DESCRIPTION:
This randomized controlled trial will include older adults aged 65 and over who have been diagnosed with medial compartment knee osteoarthritis according to the American College of Rheumatology criteria and have radiological evidence (Kellgren-Lawrence grade 2 or 3).

Eligible participants will be randomly assigned into two groups: a textured insole group and a flat insole group. Participants will wear the insoles in their daily footwear for a period of 4 weeks.

Baseline and follow-up assessments will include:

* Static and dynamic plantar pressure distribution using the Diasu® baropodometric system.
* Balance assessment using the HUR Smart Balance platform under four conditions (eyes open, eyes closed, eyes open on unstable surface, eyes closed on unstable surface).
* Functional performance tests: Timed Up and Go (TUG), 30-second Chair Stand Test, and Step Test.
* Disease-specific questionnaires: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the Knee Injury and Osteoarthritis Outcome Score (KOOS).
* Q-angle and knee proprioception measurement. Data will be analyzed to determine whether the use of textured insoles improves balance, physical performance, and plantar pressure distribution more effectively than flat insoles in older individuals with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65 and 75 years
* Diagnosed with medial compartment knee osteoarthritis
* Able to walk independently without assistive devices
* Having foot size compatible with available insole sizes
* Volunteering to participate in the study and providing informed consent

Exclusion Criteria:

* Diagnosed with neurological diseases (e.g., stroke, Parkinson's disease, multiple sclerosis)
* Diagnosed with vestibular disorders or balance problems due to inner ear issues
* Having a history of lower extremity surgery in the past year
* Severe foot deformity that prevents insole use
* Having visual impairment that is not corrected with glasses
* Currently using a walking aid (cane, walker, etc.)
* Cognitive impairment or inability to follow instructions

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in 30-Second Chair Stand Test Performance | 8 weeks
  Physical performance will be assessed using the 30-Second Chair Stand Test. The number of completed chair stands within 30 seconds will be recorded before and after the insole usage period.
Change in Timed Up and Go (TUG) Test Performance | 8 weeks
  Physical performance will be assessed using the Timed Up and Go (TUG) test. The time (in seconds) required to complete the task will be recorded before and after the insole usage period.
Change in Step Test Performance | 8 weeks
  Physical performance will be assessed using the Step Test. The number of completed steps within the allotted time will be recorded before and after the insole usage period.
Change in Static Balance Score | 8 weeks
  Static balance performance will be assessed using the HUR Smart Balance System under four conditions (eyes open, eyes closed, eyes open on unstable surface, and eyes closed on unstable surface). The static balance score will be recorded before and after the intervention.
Change in Proprioception Disturbance Score | 8 weeks
  Proprioceptive balance control will be evaluated using the proprioception disturbance score generated by the HUR Smart Balance System. Measurements will be recorded before and after the intervention.
Change in Visual Dependency Score | 8 weeks
  Visual dependency during postural tasks will be assessed using the HUR Smart Balance System under eyes open and eyes closed conditions. The visual dependency score will be recorded before and after the intervention.
Change in Left-Right Weight Distribution | 8 weeks
  Weight distribution between the left and right sides of the body will be measured using the HUR Smart Balance System during static standing. The distribution will be recorded as a percentage before and after the intervention.
Change in Peak Plantar Pressure | 8 weeks
  Peak plantar pressure (measured in kilopascals) will be assessed using the DIASU® digital baropodometric scanning system and Milletrix software. Measurements will be conducted under both barefoot and insole conditions, before and after the intervention.
Change in Plantar Contact Area | 8 weeks
  Plantar contact area (measured in square centimeters) will be assessed using the DIASU® digital baropodometric scanning system and Milletrix software. Analyses will be performed under both barefoot and insole conditions, before and after the intervention.

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data (IPD) due to the study's limited scope and ethical considerations. Data sharing might be considered in the future upon justified request and with appropriate ethical approval.

REFERENCES:
- Available data/document: Clinical Study Report — https://pubmed.ncbi.nlm.nih.gov/33946001/